CLINICAL TRIAL: NCT02802553
Title: Evaluation of an Integrated Imaging System (Smart Goggles) For In Vivo Detection of Fluorescently Labeled Lymph Nodes for Breast Cancer: A Pilot Study To Visualize Sentinel Lymph Nodes After Periareolar Injection of Indocyanine Green
Brief Title: Evaluation of an Integrated Imaging System For In Vivo Detection of Fluorescently Labeled Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE4116
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Invasive Breast Cancer
Keywords: Smart Goggles; sentinel lymph nodes; indocyanine green; Cardio-Green; Spy Elite; Quest; PDE
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Integrated Imaging Goggles (Experimental): Cardio-GreenTM (indocyanine green) peritumorally injected to breast tumor with 1 cycle. Viewed by Smart Googles and compare lesions detected by commercial FDA approved near infrared camera device (SPY Elite/Quest/PDE) in addition to those detected by gamma probe and blue dyes.
  Interventions: Device: Smart Goggle; Other: Cardio-Green; Device: SPY Elite Imaging system; Device: Quest near-infrared (NIR) Imaging system; Device: PDE Imaging system; Device: Gamma probe; Other: Blue Dyes

INTERVENTIONS:
Device: Smart Goggle — Smart Goggle is a novel stereoscopic wearable multimodal intraoperative imaging and display systems entitled Integrated Imaging Goggles for assessment of SLNs. The prototype system offers real time stereoscopic fluorescence imaging along with in vivo handheld microscopy. The investigators have found that the system can detect fluorescent targets with as low as 1.2 picomoles ICG (60 nM concentration). The hand-held microscopy module has a resolution of 25 micron. The prototype system has 2 complementary metal-oxide-semiconductor (CMOS) imaging sensors housed on a printed circuit board (PCB) with imaging lenses and emission filters optimized for ICG dye. The light source provides concurrent excitation centered at 780 nm and white light illumination with OD6 level cut-off. The Smart Goggles is a non-invasive imaging system that does not require contact with patients.
  Other Names: Integrated Imaging Goggles
Other: Cardio-Green — Indocyanine Green for Injection USP is a sterile, lyophilized green powder containing 25 mg of indocyanine green with no more than 5% sodium iodide. Indocyanine Green for Injection USP is dissolved using Sterile Water for Injection, and is to be administered intravenously.
  Other Names: Indocyanine Green
Device: SPY Elite Imaging system — Previously validated fluorescence detection system. Will be used to look at the same regions as the Smart Goggles to confirm sensitivity
Device: Quest near-infrared (NIR) Imaging system — Previously validated fluorescence detection system. Will be used to look at the same regions as the Smart Goggles to confirm sensitivity
Device: PDE Imaging system — Previously validated fluorescence detection system. Will be used to look at the same regions as the Smart Goggles to confirm sensitivity
Device: Gamma probe — Gold standard for fluorescence detection. The gamma probe and blue dyes will be used in conjunction to confirm presence of Sentinel Lymph Nodes (SLNs). The gamma probe provides non-imaging sensing data and the blue dyes provide visual signs for detection of SLNs.
Other: Blue Dyes — Gold standard for fluorescence detection. The gamma probe and blue dyes will be used in conjunction to confirm presence of Sentinel Lymph Nodes (SLNs). The gamma probe provides non-imaging sensing data and the blue dyes provide visual signs for detection of SLNs.

SUMMARY:
This is a pilot study to test and characterize the ability of the Smart Goggles system to detect fluorescently labeled sentinel lymph nodes (SLNs). Specifically, this study will test the sensitivity and specificity of the Smart Goggles to detect indocyanine green (ICG) accumulation in sentinel lymph nodes of breast cancer patients after peritumoral injection of ICG (Cardio-GreenTM), under standard-of-care application conditions.

DETAILED DESCRIPTION:
Primary Objective -Positive fluorescence signal in SLNs imaged by the Smart Goggles system.

Secondary Objectives

* Confirmation of ICG within lesions per histologic tissue exam by SLN biopsy.
* Comparison of lesions detected by the Smart Goggles vs. lesions detected using SPY/Quest/PDE vs. gold standard of gamma probe and blue dyes.

Exploratory Objectives

-Collection of preliminary data for a future, powered study for lymphatic mapping in breast cancer

Study Design This is an unpowered pilot study to determine the sensitivity of the new Smart Goggles device, for detection of ICG fluorescence in SLNs of breast cancers in a clinical setting. The investigators have chosen to examine ICG as the contrast agent and breast cancer as the clinical target, because this agent is FDA-approved and is regularly used for lymphatic mapping (skin cancers). The study team will be applying ICG for the same length of time as the standard-of-care procedures including radiotracers and blue dyes. The study involves a single visit, lasting ~3-4 hours total. Multiple SLN biopsies will be performed if multiple SLNs are identified.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with at least 1 lesion of tumor of the breast
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects who have been treated with radiation therapy on the chest.
* Has had previous sentinel lymph node biopsy
* Has a known hypersensitivity to ICG, methylene blue and 99mTc-colloid.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Binary response of the number of participants in which the Smart Goggles identifies the same Sentinel Lymph Nodes (SLN) within each participant as those identified by the gamma probe and blue dyes gold standard. | At the end of the procedure, about 50 minutes
  Agreement on 6 consecutive participants would occur less than 2% of the time by random chance (p = 0.56 = 0.016). If the two methods agree on all 6 participants, the current protocol will end successfully. However, if the two methods fail to agree on the SLN once among the first 6 participants, enrollment will continue to 25 participants or until a second failed agreement occurs.

SECONDARY OUTCOMES:
Binary response of the number of participants in which the Smart Goggles identifies the same Sentinel Lymph Nodes (SLN) within each participant as those identified by the SPY/Quest/PDE imaging systems. | At the end of the procedure, about 50 minutes
  A commercial imaging system that measures fluorescence output of ICG will be used to measure the near infrared fluorescence in vivo. Measurements are painless and involve no risk to the participant. The measurements are non-contact and recorded by a computer; each measurement is painless and takes 10 seconds. The signal is calibrated against known fluorescence standards, and the relative amount of ICG in a given measurement is interpolated from the standard curve.
Number of samples with ICG detected in biopsy tissue | At the end of the procedure, about 50 minutes
  Confirmation of ICG within lesions per histologic tissue exam by SLN biopsy.
Number of samples with lymph node detected in biopsy tissue | At the end of the procedure, about 50 minutes
  Confirmation of lymph node tissue within lesions per histologic tissue exam by SLN biopsy.
Fluorescence intensity | Typically no more than 30 minutes
  Fluorescence intensity will be compared for the removed lymph nodes between the Smart Goggles and the standard used fluorescent imaging technology. Intensity will be reported in Arbitrary units
  ·
Number of removed lymph nodes with cancer cells | At the end of the procedure, about 50 minutes
  Standard histological analyses will be performed on the biopsy specimens. Presence of absence of cancer cells in the removed lymph nodes will serve as the source of specificity.
Sensitivity as measured via the ICG accumulation curve | At the end of the procedure, about 50 minutes
  The ICG accumulation curve generated from each device (Smart Goggles vs previously validated fluorescence imaging systems), measured on the same SLN, will be used to characterize the relative sensitivity of the Smart Goggles for ICG detection in vivo.
Specificity as measured via the ICG accumulation curve | At the end of the procedure, about 50 minutes
  The ICG accumulation curve generated from each device (Smart Goggles vs previously validated fluorescence imaging systems), measured on the same SLN, will be used to characterize the relative specificity of the Smart Goggles for ICG detection in vivo.
Number of surgeons who prefer interventional device vs current near-infrared (NIR) cameras | At the end of the procedure, about 50 minutes
  Surgeons preference for using the Googles for ICG detection versus the current near-infrared NIR cameras

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Valente, DO, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States